CLINICAL TRIAL: NCT06586606
Title: A Two-Period Study to Evaluate the Effects of Multiple Oral Doses of Itraconazole on the Single Dose PK of MK-1708 in Healthy Participants
Brief Title: A Study to Evaluate the Effects of Itraconazole on MK-1708 in Healthy Participants (MK-1708-003)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1708-003; MK-1708-003 (Other: MSD)
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Period 1: MK-1708 (Experimental): Participants will receive a single oral dose of MK-1708 on Day 1.
  Interventions: Drug: MK-1708
- Period 2: MK-1708 and Itraconazole (Experimental): A washout period of at least 10 days will occur between MK-1708 dosing in Period 1 and the first itraconazole dosing in Period 2. In Period 2, participants will receive itraconazole twice daily on Day 1 and once daily on Days 2 through Day 19. Participants will also receive a single oral dose of MK-1708 on Day 4.
  Interventions: Drug: MK-1708; Drug: Itraconazole

INTERVENTIONS:
Drug: MK-1708 — Oral administration
Drug: Itraconazole — Oral administration
  Arms: Period 2: MK-1708 and Itraconazole

SUMMARY:
The goal of the study is to see what happens to levels of MK-1708 a person's body over time. Researchers will compare what happens to MK-1708 in the body when it is given with or without a medicine called itraconazole.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Is in good health before randomization
* Has a body mass index (BMI) ≥18.5 and ≤32 kg/m^2, inclusive

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* Has a history of clinically significant endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Has a history of cancer

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-10-03 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-Inf) of MK-1708 | Predose and at designated timepoints up to approximately 2 weeks postdose
  Blood samples will be collected to determine the AUC0-inf of MK-1708.
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 11 weeks
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Due to an AE | Up to approximately 11 weeks
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue study due to an AE will be reported.

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to Last Quantifiable Concentration (AUC0-Last) of MK-1708 | Predose and at designated timepoints up to approximately 2 weeks postdose
  Blood samples will be collected to determine the AUC0-last of MK-1708.
Maximum Plasma Concentration (Cmax) of MK-1708 | Predose and at designated timepoints up to approximately 2 weeks postdose
  Blood samples will be collected to determine the Cmax of MK-1708.
Time to Maximum Plasma Concentration (Tmax) of MK-1708 | Predose and at designated timepoints up to approximately 2 weeks postdose
  Blood samples will be collected to determine the Tmax of MK-1708.
Plasma Concentration at 24 Hours (C24) of MK-1708 | Predose and at designated timepoints up to 24 hours postdose
  Blood samples will be collected to determine the C24 of MK-1708.
Apparent Clearance (CL/F) of MK-1708 | Predose and at designated timepoints up to approximately 2 weeks postdose
  Blood samples will be collected to determine the CL/F of MK-1708.
Apparent Volume of Distribution During Terminal Phase (Vz/F) of MK-1708 | Predose and at designated timepoints up to approximately 2 weeks postdose
  Blood samples will be collected to determine the Vz/F of MK-1708.
Apparent Terminal Half-life (t1/2) of MK-1708 | Predose and at designated timepoints up to approximately 2 weeks postdose
  Blood samples will be collected to determine the t1/2 of MK-1708.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- QPS-MRA, LLC ( Site 0001), South Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com